CLINICAL TRIAL: NCT02677818
Title: The Relationship Between Clotting Factor VIII and Bleeding Adverse Reactions in Patients Under the Therapies of Thrombolysis, Anticoagulation and Anti-platelet
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled
Sponsor: Zhujiang Hospital (Other)
Collaborators: Guangdong Province, Department of Science and Technology (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2014-YXB-001
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Last update posted 2022-04-04 (Actual); Status verified 2021-07

CONDITIONS: Bleeding; Ischemic Stroke
Keywords: Plasma Factor VIII Levels; Ischemic stroke; Antithrombotic therapy; Bleeding
MeSH Terms: conditions — Hemorrhage; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- experimental group: The risk of bleeding adverse reactions when FVIII below the normal level.
- control group: The risk of bleeding adverse reactions when FVIII in normal level.

SUMMARY:
The purpose of this study is to determine whether Plasma Factor VIII Levels are related to the treatment of bleeding in ischemic stroke（IS）.

DETAILED DESCRIPTION:
Clear cerebral infarction patients during hospitalization, treatment process, discharge and hemorrhage occurs, the stages F VIII level change and its correlation with bleeding adverse reactions. Analysis F VIII whether belong to hemorrhage occurs independent risk factors of adverse drug reactions,as well as the feasibility of predicting bleeding occurred adverse reaction index.

ELIGIBILITY:
Inclusion Criteria:

* Guidelines prepared by the diagnostic criteria(according to the diagnostic criteria of the Fourth National Stroke Conference prepared,have been more than one times skull CT and/or MRI)was confirmed for ischemic stroke,and requires the use of antithrombotic therapy(including thrombolysis, anticoagulation, antiplatelet) patients
* Willing and able to comply with the study protocol and visits planned

Exclusion Criteria:

* At the same time the presence of other active malignancy.
* There is known brain metastases or leptomeningeal metastases
* Systemic active infection ( ie infection leads to body temperature ≥38 ℃)
* The last 4 weeks there is a need drainage ascites, pleural effusion or pericardial fluid .
* Clinically significant obstruction , pulmonary fibrosis , kidney failure , liver failure and other diseases.
* Uncontrolled diabetes.
* Severe / unstable angina, New York Heart Association (NYHA) class III or IV symptoms of congestive heart failure
* there is other reason (not the antithrombotic drugs) caused by bleeding.
* The presence of an autoimmune disease or a history of organ transplant patients require immunosuppressive therapy
* Psychiatric presence may increase the risks associated with study participation or study drug , or may interfere with the interpretation of study results
* Pregnant and lactating women
* Bleeding disorders may exist on admission
* The researchers added that the study is not appropriate to the circumstances

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The stroke patient using Anti-thrombotic drugs diagnosed by Zhujiang Hospital.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2018-01 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
The levels of FVIII are measured by enzyme-linked immuno sorbent assay. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Yong Wang, Doctor, Study Director — clinical drug trial institution
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes